CLINICAL TRIAL: NCT05071586
Title: Remotely Monitored Transcranial Direct Current Stimulation in Children With Cerebral Palsy
Brief Title: Pediatric Teleneuromodulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-0691; Protocol ver 8 5/4/2023 (Other: UW Madison); Development Pediatrics (Other: UW Madison)
Record Dates: First submitted 2021-09-13; First posted 2021-10-08 (Actual); Results first posted 2024-05-07 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-04

CONDITIONS: Cerebral Palsy (CP)
Keywords: Children with cerebral palsy; Remote transcranial direct current stimulation (tDCS); Non-invasive brain stimulation (NIBS)
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Children diagnosed with stroke/brain bleed (Experimental): Male and females aged 8 to 21 with established diagnosis of stroke/brain bleed who are US residents.
  Interventions: Device: Soterix 1x1 tDCS LTE Stimulator Device Model 1401

INTERVENTIONS:
Device: Soterix 1x1 tDCS LTE Stimulator Device Model 1401 — Participants will receive 20 minutes of 1.5 mA (Milliampere) transcranial direct current stimulation (tDCS) via Soterix 1x1 tDCS LTE Stimulator Device Model 1401 with a bilateral M1 montage.

SUMMARY:
This study will explore using remotely monitored 'active' non-invasive brain stimulation in children with cerebral palsy. Participants will receive active non-invasive brain stimulation with synchronous safety monitoring and guided instruction with laboratory staff after appropriate training. Participants will be between 8-21 years old and have a diagnosis of hemiparetic cerebral palsy with a history of a perinatal stroke or brain bleed, and can expect to be in the study for 5 days.

DETAILED DESCRIPTION:
Current exploratory single site open label unblinded trial, will assess the feasibility, tolerability, and safety of active tDCS in the home setting under caregiver, safety monitor and remote investigator supervision and direction. The study population will consist of 10 participants between ages 8 - 21 years and 365 days with hemiparetic cerebral palsy and a history of a brain bleed or stroke.

An estimated 3.6 per 1,000 births in the United States are affected by stroke or brain bleeds which can lead to Cerebral Palsy (CP), a developmental disorder associated with motor impairment. While, the majority of rehabilitation approaches focus on behavioral repetition to improve gait and upper extremity function, these therapies can require extensive practice times and extent of recovery is variable. Thus, there is a need for novel strategies which can optimize rehabilitation outcomes for this population. Brain development during childhood is characterized by heighted neuroplastic potential stressing the importance for intervention methods that harness neuroplasticity. Accordingly, several therapies are theoretically based in mechanisms of motor learning and use-dependent plasticity.

Non-invasive brain stimulation (NIBS), specifically transcranial direct current stimulation (tDCS), provides an approach for modulation of neuroplasticity that is safe, inexpensive, and portable. Furthermore, rehabilitation approaches combined with tDCS have shown promise to improve motor function recovery and quality of life after stroke in adults. Integrating the application of NIBS may allow for enhanced rehabilitation during the enhanced neuroplastic period of childhood and NIBS has demonstrated promising outcomes in increasing the rate and extent of recovery.

The Pediatric Neuromodulation laboratory has shown that in children with CP the use of tDCS is safe, feasible, and successful at modifying motor performance when in combination with other physical therapy interventions. tDCS is not currently available to subjects without taking part in the study. In this study, investigators plan to administer tDCS in the remote setting during a synchronous zoom call with trained laboratory members. To ensure the device is safely used in the home setting only during designated times, in the presence of a trained safety monitor. The safety monitor will bring the device to the session, oversee the safety of its use, and take it back to the laboratory after the session is complete.

This intervention has the potential to improve motor rehabilitation outcomes and can offer telehealth access, which may reduce treatment cost and improve access to limited access to clinic or hospital facilities. This study has the potential to set the foundation for larger clinical trials studies evaluating the efficacy of remote tDCS combined with rehabilitation interventions in children. Ultimately, this will contribute to a wider reach in improving quality of life across the lifespan in children with CP.

On Day #1 there will be a practice stimulation montage setup assessment. Before their session, a GMFCS and pediatric cognition survey will be completed with the investigative team. All participants will be asked to view instructional videos on how to perform the procedures.

Parent/child pairs will perform the assessment by walking through the steps with the guidance of the lab team member via videoconferencing. Efficiency and quality of setup data will be collected. A setup ease/comfort survey will be completed upon completion of the stimulation montage setup. Days 2-5 will consist of sham/active stimulation in the home setting under caregiver, safety monitor, and remote investigator supervision and direction. Status surveys inquiring well-being will be conducted before, during, and after stimulation as well as a Box and Blocks motor function tests. At any time the participant perceives discomfort while dosing to 1.5mA the investigators will adapt and modify the stimulation intensity.

Protocol Amendment Approved 6/7/2023: addition of an optional 6 and 12 month study visit.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 8 years 0 days and 21 years 365 days
* Children who have hemiparetic cerebral palsy with a history of perinatal brain bleed/stroke
* Receptive language function to follow two-step commands
* Able to give informed assent along with the informed consent of the legal guardian. If the participant is 18-21 (with the capacity to consent), they must be able to give informed consent.
* Intentional about representing the sub-population of children with CP who experience intellectual disability (at least 2/10 participants with mild intellectual disabilities will be recruited)
* ≥ 10 degrees of active motion at the metacarpophalangeal joint
* Children who have had surgeries, which may influence motor function e.g.- tendon transfer, will be included, yet surgical history will be documented and included in any publication within a participant characteristics table.

Exclusion Criteria:

* Inaccessibility to internet and a working computer/laptop/device.
* Implants
* Neoplasm
* Metabolic Disorders
* Epilepsy
* Seizure within two years preceding the study
* Acquired Traumatic Brain Injury
* Pregnancy
* Indwelling metal or incompatible medical devices
* Evidence of skin disease or skin abnormalities
* Botulinum toxin or Phenol block within [six-months] preceding the study
* Disorder of Cellular Migration and Proliferation

To be eligible for the optional 6-month/12-month follow-up:

* participants must have previously participated in the primary study
* have access to a reliable internet connection and a functioning computer, laptop, or mobile device.
* If participants become pregnant after participating in primary study, they may participate in the 6- and 12-month follow up sessions

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2022-12-21 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernadette Gillick, PhD, MSPT, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lench DH, Simpson E, Sutter EN, Gillick BT. Feasibility of remote transcranial direct current stimulation for pediatric cerebral palsy during the COVID-19 pandemic. Brain Stimul. 2020 Nov-Dec;13(6):1803-1804. doi: 10.1016/j.brs.2020.10.010. Epub 2020 Oct 23. No abstract available. PMID 33132132
- [Derived] Christopher P, Sutter EN, Gavioli M, Lench DH, Nytes G, Mak V, Simpson EA, Ikonomidou C, Villegas MA, Saiote C, Gillick BT. Safety, tolerability and feasibility of remotely-instructed home-based transcranial direct current stimulation in children with cerebral palsy. Brain Stimul. 2023 Sep-Oct;16(5):1325-1327. doi: 10.1016/j.brs.2023.08.024. Epub 2023 Aug 29. No abstract available. PMID 37652136
- [Derived] Simpson EA, Saiote C, Sutter E, Lench DH, Ikonomidou C, Villegas MA, Gillick BT. Remotely monitored transcranial direct current stimulation in pediatric cerebral palsy: open label trial protocol. BMC Pediatr. 2022 Sep 29;22(1):566. doi: 10.1186/s12887-022-03612-8. PMID 36175848

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Age, Customized [Count of Participants; unit: Participants]
  10 years old | 1
  13 years old | 2
  15 years old | 1
  16 years old | 4
  18 years old | 1
  19 years old | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Status/Safety Assessment
Description: Participants were asked to fill out an adverse event survey during active stimulation. Reported below are responses from the participants to the survey regardless of potential relation to stimulation.
Time Frame: Active Stimulation Sessions (20 min), 3 days total
Population: Male and females aged 8 to 21 with established diagnosis of stroke/brain bleed who are US residents.
Measure: Number; unit: number of sessions symptom reported
Units Other Than Participants: Number of Sessions
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Number analyzed (Number of Sessions) | 30
number of sessions symptom reported
  Headache | 4
  Unusual Feelings on Skin of Head | 7
  Tingling | 20
  Itchiness | 12
  Sleepiness | 7
  Difficulty paying attention | 2
  Unusual Emotions | 1
  Tooth Pain | 1
  Forgetfullness | 3
  Balance Issues | 3
  Abnormal sleep | 1

2. Primary Outcome: Change in tDCS Headgear Location
Description: To evaluate the quality of device setup, we will measure any changes or movement of the headgear. To do this, we will mark the starting and ending location of the headgear and measure the distance between the two. It will be reported if the headgear moved in any participants and the average displacement.
Time Frame: Post sessions on day 1, 2, 3, 4 , and 5
Measure: Mean (Full Range); unit: avg movement distance in inches
Units Other Than Participants: Number of Sessions
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Number analyzed (Number of Sessions) | 50
avg movement distance in inches
  Day 1 | 0.9 [0.5 to 2]
  Day 2 | 0.857 [0.25 to 2]
  Day 3 | 1.125 [0.25 to 2]
  Day 4 | 0.925 [0.2 to 1.5]
  Day 5 | 0.675 [0.2 to 1]

3. Primary Outcome: Step Difficulty Survey
Description: To evaluate the feasibility of remotely monitored-tDCS, participants were asked how difficult the setup instructions were to understand on a 5 point scale (Very easy, easy, slightly difficult, very difficult, impossible).
  Set up instruction consisted of 6 steps, participants were asked to rate the steps each day. Results are reported as overall percentage of difficulty rating over 5 days
Time Frame: Average over 5 days
Measure: Number; unit: percentage of responses
Units Other Than Participants: Number of Responses
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Number analyzed (Number of Responses) | 300
percentage of responses
  Step 1: Very Easy | 84
  Step 1: Easy | 16
  Step 1: Neural | 0
  Step 1: Difficult | 0
  Step 1: Very Difficult | 0
  Step 2: Very Easy | 74
  Step2: Easy | 20
  Step 2: Neutral | 6
  Step 2: Difficult | 0
  Step 2: Very Difficult | 0
  Step 3: Very Easy | 72
  Step 3: Easy | 20
  Step 3: Neutral | 4
  Step 3: Difficult | 4
  Step 3: Very Difficult | 0
  Step 4: Very Easy | 94
  Step 4: Easy | 6
  Step 4: Neutral | 0
  Step 4: Difficult | 0
  Step 4: Very Diffucult | 0
  Step 5: Very Easy | 94
  Step 5: Easy | 6
  Step 5: Neutral | 0
  Step 5: Difficult | 0
  Step 5: Very Difficult | 0
  Step 6: Very Easy | 60
  Step 6: Easy | 32
  Step 6: Neutral | 2
  Step 6: Difficult | 6
  Step 6: Very Difficult | 0

4. Primary Outcome: Responses to Comfort Survey
Description: To evaluate the comfort of the device, participants will be asked how comfortable was wearing the headgear on a 4 point scale(Comfortable, Slightly uncomfortable, Uncomfortable but tolerable, Very uncomfortable, and I had to remove it)
  Result reported as total over the 5 day participation in study
Time Frame: Post sessions on day 1, 2, 3, 4 , and 5
Measure: Number; unit: number of sessions when reported
Units Other Than Participants: Number of Sessions
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Number analyzed (Number of Sessions) | 50
number of sessions when reported
  Day 1: Comfortable | 9
  Day 1: Slightly uncomfortable | 1
  Day 1: Uncomfortable but tolerable | 0
  Day 1: Very uncomfortable, and I had to remove it | 0
  Day 2: Comfortable | 8
  Day 2: Slightly uncomfortable | 2
  Day 2: Uncomfortable but tolerable | 0
  Day 2: Very uncomfortable, and I had to remove it | 0
  Day 3: Comfortable | 8
  Day 3: Slightly Uncomfortable | 2
  Day 3: Uncomfortable but tolerable | 0
  Day 3: Very uncomfortable, and I had to remove it | 0
  Day 4: Comfortable | 10
  Day 4: Slightly Uncomfortable | 0
  Day 4: Uncomfortable but tolerable | 0
  Day 4: Very uncomfortable, and I had to remove it | 0
  Day 5: Comfortable | 7
  Day 5: Slightly Uncomfortable | 2
  Day 5: Uncomfortable but tolerable | 1
  Day 5: Very uncomfortable, and I had to remove it | 0

5. Secondary Outcome: Average Setup Time for Each Session
Description: To evaluate speed of device setup, time to complete montage set up will be measured and averaged among participants.
Time Frame: Pre-stimulation on day 1, 2, 3, 4 and 5
Measure: Mean (Full Range); unit: Time in seconds
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Time in seconds
  Day 1 | 530 [312 to 691]
  Day 2 | 566 [352 to 858]
  Day 3 | 622 [360 to 1008]
  Day 4 | 588 [239 to 1195]
  Day 5 | 548 [249 to 1027]

6. Secondary Outcome: Change in Box and Blocks Assessment Score
Description: To evaluate the potential change in motor function, the Box and Blocks score will be measured before and after each active session. This is a timed motor assessment, the score is the number of blocks successfully moved over a partition in one minute, a higher score indicates greater hand function. Lower scores indicate lower hand function.
  The reported outcome measure describes the change over each session in the Box and Blocks score.
  Motor function is not hypothesized to change due to the limited trials of active tDCS.
Time Frame: Post sessions on day 2, 3, 4 , and 5
Measure: Median (Standard Deviation); unit: number of blocks moved
Units Other Than Participants: number of sessions
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
Number analyzed (Participants) | 10
Number analyzed (number of sessions) | 40
number of blocks moved
  Session 2: dominant hand | 3 (2.48)
  Session 2: non- dominant hand | 0 (3.81)
  Session 3: dominant hand | 0.25 (4.75)
  Session 3: non-dominant | 1.75 (2.28)
  Session 4: dominant hand | -0.75 (4.70)
  Session 4: non-dominant hand | -2 (1.60)
  Session 5: dominant hand | 2.25 (2.40)
  Session 5: non-dominant hand | 1.5 (3.02)

ADVERSE EVENTS:
Time Frame: The adverse event survey was collected each study sham and active study visit day (day 2, 3, 4,5) before stimulation, during simulation at the 10 minute mark, and post stimulation.
Arm/Group | Children Diagnosed With Stroke/Brain Bleed
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 10/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Children Diagnosed With Stroke/Brain Bleed (N=10)
Headache (General disorders) | 4 (8)
Unusual feelings on skin of head (General disorders) | 8 (8)
Tingling (General disorders) | 9 (23)
Itching (General disorders) | 6 (17)
Sleepiness (General disorders) | 7 (14)
Difficulty paying attention (General disorders) | 6 (8)
Tooth pain (General disorders) | 1 (1)
Dizziness (General disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (3)
Forgetfulness (Psychiatric disorders) | 1 (5)
Balance (General disorders) | 1 (5)
Abnormal sleep (General disorders) | 1 (1)
Unusual emotions (Psychiatric disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-05-04): https://cdn.clinicaltrials.gov/large-docs/86/NCT05071586/Prot_SAP_002.pdf
  • Informed Consent Form (2023-04-06): https://cdn.clinicaltrials.gov/large-docs/86/NCT05071586/ICF_000.pdf